CLINICAL TRIAL: NCT05598190
Title: A577-nm Pro -Yellow Laser In Treatment of Striae Rubra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Soha Alaa Abdelaal, resident doctor atD dermatology department, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ.AST./DVA021/12/211/9/2022
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Striae Rubra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pro-Yellow laser 577 — 4 session for cases with digtal photo before and after sessions

SUMMARY:
Stretch marks or striae are common skin condition occurring in both genders, but they are more prevalent among women. These are linear dermal scars that are accompanied by epidermal atrophy. They usually occur frequently in numerous physiological and pathological conditions, such as adolescent growth, pregnancy, obesity, Cushing disease, Marfan syndrome, and long-term systemic or topical steroid use. Decreased expression of collagen and fibronectin genes has also been associated with striae.

The pro-yellow laser systems can be used in a wide range of indications such as facial erythema, facial telangiectasia, port wine stain nevus, rosacea, poikilo derma civatte, and Becker's nevus

Some of these indications are clinical lesions in the vascular pattern; some are related to the factors that trigger vascularity, such as vascular endothelial growth factor (VEGF) in etiopathogenesis

ELIGIBILITY:
Inclusion Criteria:

* .Patients diagnosed with striae rubera. .Age groups: at any age. .Sex : ( females).

  * Co-operative patient

Exclusion Criteria:

* Pregnancy .

  * Patient using drugs exacerbating stria as topical or systemic steroid, and patients using other forms of treatment for stria as topical tretinoin, emollients, glycolic acid peel and laser, because that might affect the result of our study.
  * Stria Alba.
  * Skin infection (viral, bacterial or parasitic).
  * Immunosuppressed patients or with history of malignancy or radiation therapy and chronic debilitating diseases and Cushing syndrome.
  * Hypersensitivity to light and intak of photosensitizing drugs.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
dermoscopic change of width of striae rubrae | 1 year
  dermoscopic photo for width of striae

CONTACTS AND LOCATIONS:
Locations (1):
- AZHAR University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dover JS, Rothaus K, Gold MH. Evaluation of safety and patient subjective efficacy of using radiofrequency and pulsed magnetic fields for the treatment of striae (stretch marks). J Clin Aesthet Dermatol. 2014 Sep;7(9):30-3. PMID 25276274
- [Background] Kapicioglu Y, Sarac G, Cenk H. Treatment of erythematotelangiectatic rosacea, facial erythema, and facial telangiectasia with a 577-nm pro-yellow laser: a case series. Lasers Med Sci. 2019 Feb;34(1):93-98. doi: 10.1007/s10103-018-2606-6. Epub 2018 Aug 10. PMID 30097757
- [Background] Mohamed EM, Mohamed Tawfik K, Hassan Ahmad W. Successful treatment of facial vascular skin diseases with a 577-nm pro-yellow laser. J Cosmet Dermatol. 2019 Dec;18(6):1675-1679. doi: 10.1111/jocd.12963. Epub 2019 Apr 29. PMID 31033204
- [Background] Temiz SA, Arazov S, Ataseven A, Dursun R. Treatment of Becker's nevus with 577-nm pro-yellow laser: Could it be a new treatment choice? J Cosmet Dermatol. 2021 Feb;20(2):705-706. doi: 10.1111/jocd.13882. Epub 2020 Dec 14. No abstract available. PMID 33314488